CLINICAL TRIAL: NCT01212653
Title: Effect of Anti-TNF(Alpha)Treatment on Circulating Endothelial Progenitor Cells (EPCs) and Vascular Stiffness in AS
Brief Title: Effect of Anti-TNF (Alpha) Treatment on Vascular Stiffness in Ankylosing Spondylitis (AS)
Acronym: AS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS_2010
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Ankylosing Spondylitis(AS)
Keywords: Ankylosing Spondylitis; Golimumab; Simponi; Anti-TNF alpha; EPCs; Vascular stiffness
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Golimumab (Active Comparator): In this 52-week, randomized, placebo-controlled study, patients will be randomized to receive either golimumab 50 mg monthly or matching placebo for 12 months using a 1:1 randomization procedure.
  The doctors and patients and the nurse who administer the study medication (Golimumab) will be blinded. There will be one unblinded nurse to prepare the study medication.
  Interventions: Drug: Simponi
- Pacebo-controlled (Placebo Comparator): In this 52-week, randomized, placebo-controlled study, patients will be randomized to receive either Golimumab 50 mg monthly or matching placebo for 12 months using a 1:1 randomization procedure.
  The doctors and patients and the nurse who administer the study medication (Golimumab) will be blinded. There will be one unblinded nurse to prepare the study medication.
  Interventions: Other: 0.9ml sodium chloride

INTERVENTIONS:
Drug: Simponi — Golimumab 50mg monthly
  Other Names: Golimumab
  Arms: Golimumab
Other: 0.9ml sodium chloride — 0.9ml sodium chloride
  Arms: Pacebo-controlled

SUMMARY:
1. To determine the effect of Golimumab treatment on the number and function of Endothelial Progenitor Cells (EPCs) in Ankylosing Spondylitis(AS) patients as a possible mechanism for the effect of this treatment on endothelial function.
2. To ascertain the effect of Golimumab treatment on , carotid intima-media thickness, vascular stiffness in Ankylosing Spondylitis(AS) patients as measured by pulse wave velocity (PWV) and Augmentation index (AIx).
3. To assess the clinical efficacy of Golimumab in Chinese Ankylosing Spondylitis(AS) patients according to ASAS response criteria at month 3, 6 and 12.
4. To perform cost-effectiveness and cost-utility analyses of the Golimumab in Ankylosing Spondylitis(AS) patients, using clinic-base data.

DETAILED DESCRIPTION:
This study will provide important data on the pathogenesis of vascular damage and possible mechanism by which potent anti-inflammatory treatment may reduce cardiovascular risk in Ankylosing Spondylitis(AS) patients.

Fifty patients with Ankylosing Spondylitis(AS) will be randomized to receive either Golimumab or Placebo for 12 months. Patients randomized to Placebo with worsening disease activity (failure to achieve Assessment of SpondyloArthritis international Society (ASAS20)) at week 24 will be permitted to escape to open-label Golimumab. Clinical assessment, intima-media thickness, vascular stiffness and endothelial progenitor cells will be performed at baseline, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18 years of age or older
* Fulfilled the modified New York diagnostic criteria for Ankylosing spondylitis (AS)for more than 3 months
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) ≥ 4 (0-10 point scale), Pain visual analog scale(VAS) ≥ 4 (0-10cm scale)
* Inadequate response to at least two Nonsteroidal Antiinflammatory Drugs (NASID) on highest recommended doses for 3 months or unable to receive full 3-month course because of intolerance,toxicity or contraindications
* Normal Chest X-ray within 3 months before baseline
* Purified Protein Derivative(PPD) negative, or Latent Tuberculosis (TB) patients were required therapy for Tuberculosis (TB) before or simultaneously with first dose of study agent

Exclusion Criteria:

* Complete ankylosis of the spine
* Concurrent with other inflammatory rheumatic disease
* Serious infection (treatment with IV-infective) within 2 months before randomization
* Active Tuberculosis (TB) or recent contact with a person with active Tuberculosis (TB)
* An opportunistic infection within 6 months of screening
* Known history of Hepatitis, Human Immunodeficiency Virus (HIV), Malignancy, a transplanted organ, multiple sclerosis, congestive heart failure
* Currently on systemic immunosuppressives, DMARDS (other than Methotrexate, Sulfasalazine , or Hydroxychloroquine), or Leflunomide within 4 week before first study agent
* Any previous use of Alefacept, Efalizumab, Rituximab, Golimumab or Natalizumab
* Use of cytotoxic drugs, received intra-articular, intramuscular, or intravenous corticosteroids in the past 4 weeks before screening
* Clinically significant renal disease (serum creatinine level ≥ 270µmol/L), alanine aminotransferase (ALT) ≥ 2 x upper limit of normal (ULN)
* Hemoglobin level < 8.5gm/dl, a white blood cell count < 3.5x 109/liter, a platelet count < 100x 109/liter
* Female of childbearing potential, unwilling to use adequate contraception during the study
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Effect of Golimumab treatment on the progression of subclinical atherosclerosis | Month 12
  Effect of Golimumab treatment on the progression of subclinical atherosclerosis at 12 months compared with baseline as evaluated by Intima-Media Thickness (IMT).

SECONDARY OUTCOMES:
Effect of Golimumab treatment on the changes in arterial stiffness | Month 12
  Effect of Golimumab on changes in arterial stiffness at 12 months compared with baseline as evaluated by Pulse Wave Velocity and Augmentation Index.
Changes on the number and function of Endothelial Progenitor Cells in Ankylosing Spondylitis before and after 1 year of Golimumab compared with baseline. | Month 12
  The number and function of EPCs before and after golimumab will be assessed using Wilcoxin-sign rank test
To correlate the changes in Intima-Media Thickening, Pulse Wave Velocity, Augmentation Index and Endothelial Progenitor Cells with the changes in markers of disease activity. | Month 12
  Correlation between the change in disease activity markers (BASDAI, ESR, CRP, and MRI global activity score) and the change in IMT, PWV and AIx and EPC number will be assessed using Spearman's test
Incremental cost-utility ratio of the treatment of Golimumab. | Month 12
  Utility will be assessed using the EuroQol 5D (EQ5D) and the Short-Form 36 (SF-36), at baseline and every visit.Utility is used to calculate quality-adjusted life years (QALYs). The incremental cost-utility ratio expressed as "(annual costs of golimumab treatment - annual costs of placebo treatment) / additional QALY gain by golimumab treatment" is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Derived] Tam LS, Shang Q, Kun EW, Lee KL, Yip ML, Li M, Li TK, Zhu TY, Pui MO, Li EK, Yu CM. The effects of golimumab on subclinical atherosclerosis and arterial stiffness in ankylosing spondylitis-a randomized, placebo-controlled pilot trial. Rheumatology (Oxford). 2014 Jun;53(6):1065-74. doi: 10.1093/rheumatology/ket469. PMID 24501241